CLINICAL TRIAL: NCT07132151
Title: Automated Anesthesia Systems for Painless Abortion (AAS-PA): a Multi-center, Randomized Controlled Trial
Brief Title: Reinforcement Learned Automated Anesthesia Systems During Painless Abortion
Acronym: AAS-PA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Intelligent Medical Research Center, Shenzhen United Scheme Technology Co., Ltd. (Industry)
Collaborators: Fujian Provincial Hospital (Other); Shishi Hospital (Unknown); Sichuan Provincial People's Hospital (Other); The First Affiliated Hospital of Army Medical University (Unknown); The People's Hospital of Yubei District of Chongqing city (Unknown); Peking University Shenzhen Hospital (Other); People's Hospital of Zhengzhou University (Other); Jinjiang Municipal Hospital (Shanghai Sixth People's Hospital Fujian) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZUS2025002
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Painless Abortion; Artificial Intelligence (AI); Ciprofol
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): In the test group, participants will receive anesthesia via an AI model.
  Interventions: Procedure: AI Controlled General Anesthesia
- Control group (Experimental): In the control group, anesthesia will be induced by experienced anesthesiologists.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: AI Controlled General Anesthesia — During painless abortion, anesthesia will be induced using ciprofol, and controlled by an AI model.
  Arms: Test group
Procedure: General Anesthesia — Anesthesia will be induced using ciprofol, and controlled by experienced anesthesiologists.
  Arms: Control group

SUMMARY:
This study compares the automated anesthesia systems for painless abortion (AAS-PA) with traditional anesthesia in painless abortions. It assesses intraoperative indicators (hypoxemia, injection pain, hypotension, hemodynamics, respiratory depression) and postoperative outcomes (nausea, dizziness, recovery time, satisfaction). The AAS-PA group uses AI-adjusted intravenous ciprofol based on real-time vital signs and sedation depth; the traditional group relies on manual anesthesia. The goal is to verify if AAS-PA safely manages sedation, meets painless standards, reduces adverse events, and improves experience, aiding optimized automated protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years
* ASA status Ⅰ to Ⅱ
* Diagnosed with early intrauterine pregnancy
* Body mass index (BMI) between 18 to 28 kg/m2

Exclusion Criteria:

* History of cardiac, hepatic, renal, or metabolic disorders (e.g., diabetes, hypertension, sleep apnea)
* Known allergy to opioids or ciprofloxacin components
* Cachexia
* History of substance or alcohol abuse
* ASA class III or higher
* Participation in any other drug clinical trial within the past 3 months
* Long-term use of sedative or analgesic medications
* History of neurological disorders and convulsions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2025-10-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hypoxemia | During procedure
  Hypoxemia is defined as blood oxygen saturation below 92% at any time.

SECONDARY OUTCOMES:
Area under curve of hypoxemia | During procedure
  The area where SpO2 is below 92%.
Duration of colonoscopy | During procedure
Lowest value of blood oxygen saturation | During procedure
Induction and maintenance doses of anesthesia | During procedure
  Doses are recorded in mg/kg/h. The induction period is defined as the interval from the start of anesthesia to the first BIS value below 60. The maintenance period is defined as the interval from the first BIS value below 60 to the end of the drug infusion.
Ciprofol related adverse reactions | During procedure
  Included sinus bradycardia, dizziness
Induction time | During procedure
  The time interval from the start of drug administration to the first BIS ≤ 1.
Complete recovery time | During procedure
  Time interval from cessation of anesthetic agents to BIS > 80.
Incidence of hypotension | During procedure
  Systolic blood pressure < 90 mmHg or a 30% decrease from baseline lasting longer than 2 minutes.
Counts of body movement | During procedure
Dose of norepinephrine | During procedure

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Jinjiang Municipal Hospital (Shanghai Sixth People's Hospital Fujian), Jinjiang, Fujian
  - Shishi Hospital, Quanzhou, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Army Medical University, Chongqing
  - The People's Hospital of Yubei District of Chongqing city, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided